CLINICAL TRIAL: NCT01805453
Title: Angiotensin II Receptor Blockers, Steroids and Radiotherapy in Glioblastoma- A Randomized Multicenter Trial
Brief Title: Angiotensin II Receptor Blockers, Steroids and Radiotherapy in Glioblastoma
Acronym: ASTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ANOCEF (french association of neuro-oncologists) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P120105; 2012-004536-34 (EudraCT Number)
Record Dates: First submitted 2013-02-25; First posted 2013-03-06 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Newly-diagnosed Glioblastoma
Keywords: Glioblastoma; Angiotensin-II inhibitors; Losartan; steroids; Radiotherapy; Edema; Randomized trial
MeSH Terms: conditions — Glioblastoma; Edema | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Losartan (Active Comparator): Arm A: Standard of care (Radiotherapy with concomitant temozolomide followed by monthly cures of temozolomide ) + Losartan 50mg*2/day until the halting for any reason
  Interventions: Drug: Losartan
- Arm B: Placebo (Placebo Comparator): Arm B: Standard of care (Radiotherapy with concomitant temozolomide followed by monthly cures of temozolomide + Placebo 2/day until the halting for any reason
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Standard of care (Radiotherapy with concomitant temozolomide followed by monthly cures of temozolomide ) + Losartan or placebo (Arm A or B) 50mg*2/day until the halting for any reason
  Arms: Arm A: Losartan
Drug: Placebo — Standard of care (Radiotherapy with concomitant temozolomide followed by monthly cures of temozolomide + Placebo 2/day until the halting for any reason
  Arms: Arm B: Placebo

SUMMARY:
To assess the efficacy of an Angiotensin-II inhibitor (Losartan) to reduce peritumoral edema in newly diagnosed glioblastoma patients.

DETAILED DESCRIPTION:
Multicentre, randomized (1:1), double blinded trial:- Arm A: Standard of care (Radiotherapy with concomitant temozolomide followed by monthly cures of temozolomide ) + Losartan 50mg*2/day until the halting for any reason - Arm B: Standard of care (Radiotherapy with concomitant temozolomide followed by monthly cures of temozolomide + Placebo 2/day until the halting for any reason.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Histologically confirmed glioblastoma (Grade 4 WHO)
* patients eligible for radiotherapy and concomitant Temozolomide
* KPS ≥ 50%
* Adequate hematologic, liver and renal functions

Exclusion Criteria:

* Patients unable to undergo an MRI with contrast
* Patients without any residual tumor left on the screening MRI of both flair and contrast-enhanced lesions complete surgical resection)
* Any prior treatment of glioblastoma including any local therapy (immunotherapy, Gliadel wafers, …..) during or after surgical resection
* Any on-going treatment for high blood pressure at time of inclusion, whatever the therapeutic class of drugs
* Systolic blood pressure <110 mmHg.
* relative or definite contra-indication to Losartan:
* Pregnant or breast feeding women; Women with an intact uterus (unless amenorrhoeic for the last 24 months) not using effective means of contraception
* Non-affiliation to the "sécurité sociale"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Steroid dosage required to control brain edema on the last day of radiotherapy in each arm | Up to Day 42+ 1 month

SECONDARY OUTCOMES:
Steroids dosage 1 month after the end of RT | Day 42+ 1 month
Assessment of cerebral edema on MRI | Day -28 at -13, Day 42, Day 42+1 month
Tolerance (NCI-CTCAE v3.0) | up to day42 +1 month + 7 days
  To be reported according to NCI/CTC version 3.0 (adverse events)
Blood pressure | Day -10 at -7, Day0, 42, Day 42+1month
HbA1C | Day -10 at -7, D42, Day 42+1month
glycemia | Day -10 at -7, Day14, 28, 42, Day 42+1month
body weight | Day -10 at -7, Day42, Day 42+1month
side-effects of steroids | up to day42 +1 month
Executive functions ( " Moca test ") | Day-10 at -7, Day 42, Day 42+1 month
Quality of life (EORTC) | Day-10 at -7, Day 42, Day 42+1 month
Progression free survival | up to 24 months
Overall survival | up to 24 months
Survival | at 1 year, 2 year
Performance status (KPS) at the end, 1 month , and 2 months after the end of RT | at the end, 1 month, and 2 months after the end of RT

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CARPENTIER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Neurology Department - Avicenne Hospital, Bobigny, France

REFERENCES:
- [Derived] Ursu R, Thomas L, Psimaras D, Chinot O, Le Rhun E, Ricard D, Charissoux M, Cuzzubbo S, Sejalon F, Quillien V, Hoang-Xuan K, Ducray F, Portal JJ, Tibi A, Mandonnet E, Levy-Piedbois C, Vicaut E, Carpentier AF. Angiotensin II receptor blockers, steroids and radiotherapy in glioblastoma-a randomised multicentre trial (ASTER trial). An ANOCEF study. Eur J Cancer. 2019 Mar;109:129-136. doi: 10.1016/j.ejca.2018.12.025. Epub 2019 Feb 1. PMID 30716716